CLINICAL TRIAL: NCT05645809
Title: A Multicenter, Randomized, Single-blinded, Active Controlled, Non-inferiority, Post Marketing Clinical Trial to Evaluate the Safety and Efficacy of MONOFIX® PGCL Suture Compared to Quill MonodermTM Suture in Laparoscopic Surgery
Brief Title: Clinical Trial to Evaluate the Safety and Efficacy of MONOFIX® PGCL Suture in Laparoscopic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Samyang Biopharmaceuticals Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: MF_PGCL_401
Record Dates: First submitted 2022-11-17; First posted 2022-12-12 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: Laparoscopic Hysterectomy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MONOFIX® PGCL (Experimental): An absorbable suture
  Interventions: Device: MONOFIX® PGCL
- Quill Monoderm™ (Active Comparator): An absorbable suture
  Interventions: Device: Quill Monoderm™

INTERVENTIONS:
Device: MONOFIX® PGCL — An absorbable suture made of polyglycapron (PGCL) used for soft tissue suture.
  Arms: MONOFIX® PGCL
Device: Quill Monoderm™ — An absorbable suture made of polyglactin used for soft tissue suture.
  Arms: Quill Monoderm™

SUMMARY:
Clinical Trial to Evaluate the Safety and Efficacy of MONOFIX® PGCL Suture Compared to Quill MonodermTM Suture in Laparoscopic Surgery

ELIGIBILITY:
Inclusion Criteria:

1. Patients scheduled for hysterectomy by laparoscopic surgery

* Patients who are scheduled to undergo hysterectomy after being diagnosed with benign tumors in the uterus, including uterine myoma, according to the medical judgment of the investigator
* Laparoscopic surgery includes general laparoscopic surgery and robotic surgery.)

Exclusion Criteria:

1. Patients with contaminated wounds
2. Diseases that may affect wound healing
3. When gynecological malignancy or intra-abdominal metastasis is confirmed at the time of enrollment

Min Age: 19 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2022-11-03 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Time used for suturing the surgical site during laparoscopic hysterectomy | 0Day
  Time used from when the first suture is started to when the last suture is finished and the suture is cut

CONTACTS AND LOCATIONS:
Overall Officials: Jinhwa Hong, Principal Investigator — Korea University Guro Hospital
Locations (1):
- Korea University Guro Hospital, Seoul, South Korea